CLINICAL TRIAL: NCT00219076
Title: A Six-week, Randomized, Double-blind, Parallel-group, Multicenter Study to Evaluate the Safety and Efficacy of the Combination of Aliskiren 150 mg and Amlodipine 5 mg Compared to Amlodipine 5 mg and 10 mg in Hypertensive Patients Not Adequately Responsive to Amlodipine 5 mg
Brief Title: A Clinical Study to Evaluate the Safety and Efficacy of the Combination of Aliskiren and Amlodipine in Hypertensive Non Responders Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CSPP100A2305
Record Dates: First submitted 2005-09-12; First posted 2005-09-22 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Hypertension
Keywords: Hypertension, aliskiren, blood pressure, amlodipine
MeSH Terms: conditions — Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: aliskiren

SUMMARY:
To evaluate the blood pressure lowering effect and safety of aliskiren 150 mg used in combination with amlodipine 5 mg in patients with essential hypertension not adequately responsive to amlodipine 5 mg.

ELIGIBILITY:
Inclusion Criteria

* Patients with essential hypertension
* Patients who are eligible and able to participate in the study Exclusion Criteria
* Severe hypertension
* History or evidence of a secondary form of hypertension
* History of Hypertensive encephalopathy or cerebrovascular accident. Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504
Dates: Start 2005-02; Primary Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean sitting diastolic blood pressure after 6 weeks

SECONDARY OUTCOMES:
Change from baseline in mean sitting systolic blood pressure after 6 weeks
Mean sitting diastolic blood pressure < 90 mmHg or a reduction of > 10 mmHg after 6 weeks
Achieve mean sitting blood pressure target of < 140/90 mmHg after 6 weeks
Change from baseline in standing diastolic blood pressure after 6 weeks
Change from baseline in standing systolic blood pressure after 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Novartis Pharmaceuticals, East Hanover, New Jersey, United States
- Investigative Centers, Germany